CLINICAL TRIAL: NCT02277990
Title: Cardiac Implantable Electronic Device (CIED) Antibiotic Envelope Infection Prevention Trial
Brief Title: World-wide Randomized Antibiotic Envelope Infection Prevention Trial
Acronym: WRAP-IT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WRAP-IT
Record Dates: First submitted 2014-10-22; First posted 2014-10-29 (Estimated); Results first posted 2019-10-24 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: CIED Related Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TYRX™ envelope (Active Comparator): The Medtronic TYRX™ Absorbable Antibacterial Envelope is an absorbable sterile prosthesis designed to hold a pacemaker pulse generator or defibrillator to create a stable environment when implanted in the body. The purpose of the absorbable coating is to act as a carrier for the antimicrobial agents.
  Interventions: Device: TYRX™ Absorbable Antibacterial Envelope
- Control (No Intervention): No TYRX™ envelope, bare CIED

INTERVENTIONS:
Device: TYRX™ Absorbable Antibacterial Envelope
  Arms: TYRX™ envelope

SUMMARY:
Medtronic , Inc. is sponsoring the World-wide Randomized Antibiotic Envelope Infection Prevention Trial (WRAP-IT), a randomized, prospective, multi-center, single blinded, post-market, interventional clinical study. This study will evaluate the ability of the TYRX™ envelope to reduce major Cardiac Implantable Electronic Device (CIED) infections through 12-months post-procedure following CIED generator replacement, upgrade, revision, or de novo cardiac resynchronization therapy defibrillator (CRT-D) implant. Additionally, this large device study provides the unique opportunity to prospectively characterize the performance of Medtronic's lead monitoring features in subjects whose CIED system includes a transvenous right ventricular (RV) defibrillation lead. Finally, the WRAP-IT study will serve as a post-approval study for those geographies requiring a post-approval study of the TYRX™ envelope.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing to sign and date the study patient informed consent (PIC) form
* Patient is at least 18 years of age and meets age requirements per local law
* Patient is planned to undergo at least one of the following:

  a. Patient has existing cardiac implantable electronic device (CIED) and is undergoing implantable pulse generator (IPG) (including cardiac resynchronization therapy pacemaker [CRT-P]), implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D) replacement or upgrade with a new Medtronic generator

  i. Subjects planned to have leads added, or extracted and added for upgrades can be enrolled OR

  b. Patient will undergo a de novo Medtronic CRT-D system implant per approved indications

OR

c. Patient has existing study eligible Medtronic CIED in which the pocket was not accessed within the last 365 days, and is undergoing pocket or lead revision

* Willing to provide the contact information for the physician who provides followup for his/her CIED
* Willing and able to comply with scheduled follow-up and study related activities

Exclusion Criteria:

* Known allergy to minocycline or rifampin or their derivatives, or any other known contraindications to implantation of the TYRX envelope.
* Current therapy with chronic oral immunosuppressive agents or ≥ 20mg/day of Prednisone or equivalent.
* Hemodialysis or peritoneal dialysis.
* Prior Cardiac transplantation or existing Ventricular Assist Device (VAD).
* Require long-term vascular access for any reason.
* Prior history of a CIED infection, other prosthetic device infection, or endovascular infection, including endocarditis, in the past 12 months.
* Physical, clinical, or laboratory signs or symptoms consistent with an active infection (including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia)
* Systemic lupus erythematous, because minocycline has been reported to aggravate this condition
* Female patient who is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within 7 days prior to device procedure
* Participation in another study that may confound the results of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from the Medtronic study manager.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7075 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wilkoff, MD, Study Chair — The Cleveland Clinic; Khaldoun Tarakji, MD, Principal Investigator — The Cleveland Clinic
Locations (181):
- United States (120):
  - Alaska Heart Institute, Anchorage, Alaska
  - Tri-City Cardiology Consultants, Mesa, Arizona
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Chula Vista Cardiac Center, Chula Vista, California
  - Cardiovascular Consultants Heart Center, Fresno, California
  - UCSD Medical Center, La Jolla, California
  - Eisenhower Desert Cardiology Center, Rancho Mirage, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Stanford Hospital & Clinics, Stanford, California
  - Saint Joseph's Medical Center, Stockton, California
  - Penrose St. Francis Hospital, Colorado Springs, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - SCL Physicians Heart Institute of Colorado, Lafayette, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Florida Electrophysiology Associates, Atlantis, Florida
  - Clearwater Cardiovascular & Interventional Consultants, Clearwater, Florida
  - The Cardiac & Vascular Institute, Gainesville, Florida
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - Kootenai Heart Clinics Northwest, Coeur d'Alene, Idaho
  - NorthShore University Health System, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Prairie Education & Research Cooperative (Springfield IL), Springfield, Illinois
  - Saint Vincent Medical Group, Indianapolis, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - The University Kansas Medical Center Research Institute Inc, Kansas City, Kansas
  - Lexington Cardiac Research Foundation, Lexington, Kentucky
  - Norton Cardiovascular Associates, Louisville, Kentucky
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Advanced Cardiovascular Specialists, Shreveport, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - MedStar Health Research Institute, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Delmarva Heart Research Foundation Inc, Salisbury, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - DLP Marquette Physicians Practices Inc, Marquette, Michigan
  - Upper Michigan Cardiovascular Associates PC, Marquette, Michigan
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Great Lakes Heart and Vascular Institute PC, Saint Joseph, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Hattiesburg Clinic/ Forrest General, Hattiesburg, Mississippi
  - Mid America Heart Institute (MAHI), Kansas City, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Saint Anthonys Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Englewood Hospital & Medical Center, Englewood, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Saint Joseph's Hospital Health Center, Liverpool, New York
  - Cornell University Medical Center, New York, New York
  - Mount Sinai Saint Luke's Hospital, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - NYU, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Westchester Medical Center, Valhalla, New York
  - Asheville Cardiology Associate PA, Asheville, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Raleigh Cardiology Associates, Raleigh, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences / Baptist Medical Center / North Carolina Baptist Hospital, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Northeast Ohio Cardiovascular Specialists, Akron, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Saint Elizabeth Health Center, Poland, Ohio
  - Mount Carmel East, Westerville, Ohio
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - University of Oklahoma Health Science Center (OUHSC), Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Legacy Medical Group, Portland, Oregon
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Providence Health & Services, Portland, Oregon
  - Lehigh Valley Hospital Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Hospital, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Doylestown Cardiology Associates - VIAA, Doylestown, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Hamot, Erie, Pennsylvania
  - Saint Mary Medical Center (Langhorne PA), Newtown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - The Miriam Hospital, East Providence, Rhode Island
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Jackson Clinic, Jackson, Tennessee
  - Wellmont CVA Heart Institute, Kingsport, Tennessee
  - Centennial Heart Cardiovascular Consultants LLC, Nashville, Tennessee
  - Saint Thomas Research Institute, Nashville, Tennessee
  - Amarillo Heart Group, Amarillo, Texas
  - Cardiology Associates of Corpus Christi, Corpus Christi, Texas
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - North Texas Heart Center, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Longview Regional Medical Center, Longview, Texas
  - Baylor Research Institute, Plano, Texas
  - Scott & White Health Science Ctr, Temple, Texas
  - EP Heart LLC, The Woodlands, Texas
  - The University of Vermont Medical Center Inc, Burlington, Vermont
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Inc., Green Bay, Wisconsin
- Universitätsklinikum Krems, Krems, Austria
- Belgium (3):
  - Universitair Ziekenhuis Brussel, Brussels
  - Ziekenhuis Oost Limburg - Campus St.-Jan, Genk
  - Centre Hospitalier Regional de la Citadelle, Liège
- Canada (4):
  - Saint Paul's Hospital (Vancouver BC), Vancouver, British Columbia
  - Hamilton General Hospital / Hamilton Health Sciences, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec
- Hospital San Juan de Dios, Santiago, Chile
- China (2):
  - Grantham Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
- Rigshospitalet, Copenhagen, Denmark
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turun Yliopistollinen keskussairaala, Turku
- France (5):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Hôpital de la Timone - Centre Hospitalier Universitaire de Marseille, Marseille
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU Hôpiteaux de Rouen - Hôpital Charles Nicolle, Rouen
  - Centre Hospitalier Universitaire Saint Étienne - Hôpital Nord, Saint-Priest-en-Jarez
- Germany (2):
  - Universitäts-Herz-Zentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Universitätsmedizin Rostock, Rostock
- Greece (3):
  - University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - Onassis Cardiac Surgery Center, Kallithea
- Israel (2):
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (4):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Presidio Ospedaliero Sant'Anna, Como
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Malaysia (3):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Institut Jantung Negara - National Heart Institute, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- Helse Bergen HF - Haukeland Universitetssjukehus, Bergen, Norway
- Poland (2):
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Szpital Kliniczny Przemienienia Panskiego, Poznan
- Portugal (2):
  - Hospital de Santa Maria-Centro Hospitalar Lisboa Norte, EPE, Lisbon
  - Centro Hospitalar do Porto, Porto
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia
- Singapore (2):
  - Changi General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
- Slovakia (3):
  - Stredoslovensky ustav srdcovych a cievnych chorob a.s, Banská Bystrica
  - Narodny ustav srdcovych a cievnych chorob, a.s. (NUSCH), Bratislava
  - Vychodoslovensky ustav srdcovych a cievnych chorob, a.s., Košice
- Spain (4):
  - Hospital Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitari Bellvitge, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
- Sweden (4):
  - Alingsås Lasarett, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Stockholm
  - Sjukhuset i Varberg, Varberg
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Cardiocentro Ticino, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
- United Kingdom (4):
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Royal Brompton & Harefield NHS Foundation Trust - Harefield Hospital, London
  - Central Manchester University Hospitals NHS - Manchester Royal Infirmary, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Poole JE, Swerdlow CD, Tarakji KG, Mittal S, Ellenbogen KA, Greenspon AJ, Kennergren C, Philbert BT, Moore J, Jones RC, Schaller RD, Hansalia R, Simmers T, Mihalcz A, DeBus B, Lexcen DR, Gunderson B, Wilkoff BL. Clinical performance of implantable cardioverter-defibrillator lead monitoring diagnostics. Heart Rhythm. 2022 Mar;19(3):363-371. doi: 10.1016/j.hrthm.2021.10.032. Epub 2021 Nov 9. PMID 34767985
- [Derived] Sohail MR, Corey GR, Wilkoff BL, Poole JE, Mittal S, Kennergren C, Greenspon AJ, Cheng A, Lande JD, Lexcen DR, Tarakji KG. Clinical Presentation, Timing, and Microbiology of CIED Infections: An Analysis of the WRAP-IT Trial. JACC Clin Electrophysiol. 2021 Jan;7(1):50-61. doi: 10.1016/j.jacep.2020.07.021. Epub 2020 Oct 28. PMID 33478712
- [Derived] Wilkoff BL, Boriani G, Mittal S, Poole JE, Kennergren C, Corey GR, Krahn AD, Schloss EJ, Gallastegui JL, Pickett RA, Evonich RF, Roark SF, Sorrentino DM, Sholevar DP, Cronin EM, Berman BJ, Riggio DW, Khan HH, Silver MT, Collier J, Eldadah Z, Holbrook R, Lande JD, Lexcen DR, Seshadri S, Tarakji KG. Cost-Effectiveness of an Antibacterial Envelope for Cardiac Implantable Electronic Device Infection Prevention in the US Healthcare System From the WRAP-IT Trial. Circ Arrhythm Electrophysiol. 2020 Oct;13(10):e008503. doi: 10.1161/CIRCEP.120.008503. Epub 2020 Sep 11. PMID 32915063
- [Derived] Wilkoff BL, Boriani G, Mittal S, Poole JE, Kennergren C, Corey GR, Love JC, Augostini R, Faerestrand S, Wiggins SS, Healey JS, Holbrook R, Lande JD, Lexcen DR, Willey S, Tarakji KG; WRAP-IT Investigators. Impact of Cardiac Implantable Electronic Device Infection: A Clinical and Economic Analysis of the WRAP-IT Trial. Circ Arrhythm Electrophysiol. 2020 May;13(5):e008280. doi: 10.1161/CIRCEP.119.008280. Epub 2020 Apr 12. PMID 32281393
- [Derived] Mittal S, Wilkoff BL, Kennergren C, Poole JE, Corey R, Bracke FA, Curnis A, Addo K, Martinez-Arraras J, Issa ZF, Redpath C, Moubarak J, Khelae SK, Boersma LVA, Korantzopoulos P, Krueger J, Lande JD, Morss GM, Seshadri S, Tarakji KG. The World-wide Randomized Antibiotic Envelope Infection Prevention (WRAP-IT) trial: Long-term follow-up. Heart Rhythm. 2020 Jul;17(7):1115-1122. doi: 10.1016/j.hrthm.2020.02.011. Epub 2020 Feb 19. PMID 32087357
- [Derived] Tarakji KG, Mittal S, Kennergren C, Corey R, Poole JE, Schloss E, Gallastegui J, Pickett RA, Evonich R, Philippon F, McComb JM, Roark SF, Sorrentino D, Sholevar D, Cronin E, Berman B, Riggio D, Biffi M, Khan H, Silver MT, Collier J, Eldadah Z, Wright DJ, Lande JD, Lexcen DR, Cheng A, Wilkoff BL; WRAP-IT Investigators. Antibacterial Envelope to Prevent Cardiac Implantable Device Infection. N Engl J Med. 2019 May 16;380(20):1895-1905. doi: 10.1056/NEJMoa1901111. Epub 2019 Mar 17. PMID 30883056

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 92 total patients that were enrolled into the study, but not randomized. After enrollment, but prior to randomization, 2 patients died, 31 patients were found to not meet eligibility criteria, 50 patients withdrew, 1 investigator withdrew the patient and 8 patients had an other or unknown reason for not being randomized.
Groups:
- TYRX Envelope: The Medtronic TYRX Absorbable Antibacterial Envelope is an absorbable sterile prosthesis designed to hold a pacemaker pulse generator or defibrillator to create a stable environment when implanted in the body. The purpose of the absorbable coating is to act as a carrier for the antimicrobial agents.
  TYRX Absorbable Antibacterial Envelope
- Control: No TYRX envelope, bare CIED
Period: Overall Study
Arm/Group | TYRX Envelope | Control
Started (Randomized: Per the study protocol, only randomized subjects are included in the analysis cohort.) | 3495 | 3488
Completed (Definition of completed is that subject was followed to 12 months) | 3129 | 3112
Not Completed | 366 | 376
Not completed — Death | 170 | 188
Not completed — Withdrawal by Subject | 64 | 53
Not completed — Physician Decision | 40 | 34
Not completed — Lost to Follow-up | 66 | 69
Not completed — Had other reason | 26 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TYRX Envelope | Control | Total
Number analyzed (Participants) | 3495 | 3488 | 6983
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 8 participants did not complete a baseline characteristics form
  years
    number analyzed (Participants) | 3490 | 3485 | 6975
    (all) | 70.0 (12.6) | 70.1 (12.4) | 70.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 997 | 976 | 1973
  Male | 2498 | 2512 | 5010
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 8 participants did not complete a baseline characteristics form
  Participants
    number analyzed (Participants) | 3490 | 3485 | 6975
    American Indian or Alaska Native | 8 | 4 | 12
    Asian | 97 | 91 | 188
    Native Hawaiian or Other Pacific Islander | 9 | 7 | 16
    Black or African American | 202 | 207 | 409
    White | 2698 | 2691 | 5389
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 476 | 485 | 961
Region of Enrollment [Number; unit: participants]
  Singapore | 11 | 8 | 19
  United States | 2440 | 2441 | 4881
  Malaysia | 42 | 41 | 83
  Portugal | 20 | 17 | 37
  Greece | 45 | 43 | 88
  Saudi Arabia | 11 | 10 | 21
  Austria | 29 | 29 | 58
  Netherlands | 70 | 69 | 139
  Sweden | 45 | 47 | 92
  China | 18 | 19 | 37
  Poland | 18 | 16 | 34
  Slovakia | 29 | 31 | 60
  Chile | 2 | 3 | 5
  France | 94 | 94 | 188
  United Kingdom | 135 | 141 | 276
  Switzerland | 30 | 33 | 63
  Spain | 52 | 48 | 100
  Canada | 131 | 131 | 262
  Belgium | 36 | 35 | 71
  Norway | 32 | 32 | 64
  Finland | 24 | 23 | 47
  Denmark | 34 | 36 | 70
  Italy | 88 | 86 | 174
  Israel | 47 | 44 | 91
  Germany | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Kaplan-Meier Estimate of Major CIED Infection Rate
Description: CIED infections are defined as (1) superficial cellulitis in the region of the CIED pocket with wound dehiscence, erosion, or purulent drainage, (2) deep incisional or organ/space (generator pocket) surgical site infection that meets the Centers for Disease Control and Prevention criteria, independent from time of surgery, (3) persistent bacteremia, or (4) endocarditis.
  Major CIED infections are defined as a CIED infection resulting in one or more of the following:
  * CIED system removal
  * Any invasive procedure (e.g. pocket opened) without system removal
  * Treatment with antibiotic therapy if the subject is not a candidate for system removal and infection recurrence after completion of antibiotic therapy or evidence of deep infection with wound dehiscence, erosion, or purulent drainage
  * Death
Time Frame: Implant to 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TYRX Envelope | Control
Number analyzed (Participants) | 3495 | 3488
Percentage of subjects | 0.7 [0.5 to 1.1] | 1.2 [0.9 to 1.7]
Statistical Analysis 1: Comparison: TYRX Envelope vs Control; Test type: Superiority; p = 0.0406, Regression, Cox — The 0.05 critical value for assessing the primary endpoint was adjusted to 0.0488, to account for a planned interim analysis; The Cox regression was stratified according to device type (pacemaker or CRT-P vs. ICD or CRT-D); Hazard Ratio (HR) = 0.60, 95.12% CI 2-sided [0.36 to 0.98]

2. Secondary Outcome: 12 Month Kaplan-Meier Estimate of Major or Minor CIED Infection
Description: Major CIED infections are defined above. Minor CIED infections are defined as CIED infections that do not meet the definition of a major CIED infection
Time Frame: Implant to 12 months
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TYRX Envelope | Control
Number analyzed (Participants) | 3495 | 3488
Percentage of subjects | 1.4 [1.1 to 2.0] | 2.2 [1.8 to 2.8]
Statistical Analysis 1: Comparison: TYRX Envelope vs Control; Test type: Superiority; p = 0.0248, Regression, Cox; Hazard Ratio (HR) = 0.67, 95.12% CI 2-sided [0.47 to 0.96]

3. Secondary Outcome: 12 Month Kaplan-Meier Estimate of a CIED Procedure Related or System Related Complication
Description: * A CIED system related event is defined as an adverse event related to the CIED system which includes the device, leads, implant tool(s), programmer, or TYRX envelope (if applicable)
  * A CIED procedure related event is defined as an adverse event that occurs due to any procedure related to the implantation or surgical modification of the system including the TYRX envelope (if applicable)
  * A procedure or system related complication is defined as an adverse event related to a CIED procedure or the CIED system that results in at least one of the following:
  Death,Termination of significant device function, Invasive intervention
Time Frame: Implant to 12 months
Population: Per the Statistical Analysis Plan, the statistical inference for this objective was based on the As-Treated cohort instead of the Intention-to-Treat cohort. Per the cohort definition, subjects are analyzed based on the treatment (envelope or no envelope) and the device class (low or high power) that was actually received.
Measure: Number; unit: Percentage of subjects
Arm/Group | TYRX Envelope | Control
Number analyzed (Participants) | 3396 | 3507
Percentage of subjects | 6.0 | 6.9
Statistical Analysis 1: Comparison: TYRX Envelope vs Control; Test type: Non-Inferiority — The non-inferiority test was performed on the as-treated cohort, per the statistical analysis plan. The non-inferiority margin for the hazard ratio was 1.33 (i.e., the hazard ratio for complications in the envelope group vs. the control group must be significantly lower than 1.33); p < 0.01, Regression, Cox; Hazard Ratio (HR) = 0.93, 95.12% CI 2-sided [0.77 to 1.12]

4. Secondary Outcome: Kaplan-Meier Estimate of a Major Infection Throughout Follow-up
Description: as for outcome 1
Time Frame: Throughout study follow-up Kaplan-Meier Estimate is at 36 Months
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | TYRX Envelope | Control
Number analyzed (Participants) | 3495 | 3488
Percentage of subjects | 1.3 [0.09 to 2.0] | 1.9 [1.4 to 2.6]
Statistical Analysis 1: Comparison: TYRX Envelope vs Control; Test type: Superiority; p = 0.0402, Regression, Cox; Hazard Ratio (HR) = 0.63, 95.12% CI 2-sided [0.40 to 0.98]

ADVERSE EVENTS:
Time Frame: Assessed from baseline visit to 36-month follow-up visit
Arm/Group | TYRX Envelope | Control
All-Cause Mortality (participants affected / at risk) | 349/3495 | 365/3488
Serious Adverse Events (participants affected / at risk) | 1553/3495 | 1548/3488
Other Adverse Events (participants affected / at risk) | 286/3495 | 221/3488
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TYRX Envelope (N=3495) | Control (N=3488)
Anaemia (Blood and lymphatic system disorders) | 28 | 26
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 2 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 9 | 3
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 10
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 4
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 32 | 35
Angina pectoris (Cardiac disorders) | 20 | 29
Angina unstable (Cardiac disorders) | 15 | 10
Aortic valve disease (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 4 | 0
Aortic valve stenosis (Cardiac disorders) | 3 | 3
Arrhythmia (Cardiac disorders) | 5 | 8
Arrhythmia supraventricular (Cardiac disorders) | 2 | 4
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 127 | 136
Atrial flutter (Cardiac disorders) | 21 | 18
Atrial tachycardia (Cardiac disorders) | 6 | 6
Atrial thrombosis (Cardiac disorders) | 2 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 36 | 23
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 2
Cardiac failure (Cardiac disorders) | 131 | 131
Cardiac failure acute (Cardiac disorders) | 35 | 48
Cardiac failure chronic (Cardiac disorders) | 14 | 26
Cardiac failure congestive (Cardiac disorders) | 186 | 200
Cardiac perforation (Cardiac disorders) | 1 | 1
Cardiac tamponade (Cardiac disorders) | 3 | 5
Cardiac valve disease (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 13 | 10
Cardiogenic shock (Cardiac disorders) | 18 | 15
Cardiomyopathy (Cardiac disorders) | 19 | 15
Cardiomyopathy alcoholic (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 2 | 6
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Chronic left ventricular failure (Cardiac disorders) | 5 | 4
Congestive cardiomyopathy (Cardiac disorders) | 0 | 6
Coronary artery disease (Cardiac disorders) | 32 | 32
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 3
Coronary artery stenosis (Cardiac disorders) | 1 | 3
Hypertensive heart disease (Cardiac disorders) | 0 | 2
Intracardiac thrombus (Cardiac disorders) | 0 | 6
Ischaemic cardiomyopathy (Cardiac disorders) | 9 | 18
Left ventricular dysfunction (Cardiac disorders) | 4 | 3
Left ventricular failure (Cardiac disorders) | 3 | 4
Mitral valve disease (Cardiac disorders) | 3 | 1
Mitral valve incompetence (Cardiac disorders) | 8 | 11
Mitral valve stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 11 | 10
Myocardial ischaemia (Cardiac disorders) | 3 | 3
Palpitations (Cardiac disorders) | 4 | 3
Pericardial effusion (Cardiac disorders) | 11 | 7
Pulseless electrical activity (Cardiac disorders) | 4 | 1
Rheumatic heart disease (Cardiac disorders) | 0 | 1
Right atrial dilatation (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 2 | 2
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 5 | 8
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 9 | 6
Torsade de pointes (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 4 | 1
Ventricular arrhythmia (Cardiac disorders) | 19 | 10
Ventricular extrasystoles (Cardiac disorders) | 2 | 7
Ventricular fibrillation (Cardiac disorders) | 22 | 26
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 92 | 92
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Congenital aortic valve stenosis (Congenital, familial and genetic disorders) | 0 | 1
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Myotonic dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 4
Vertigo labyrinthine (Ear and labyrinth disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 3 | 0
Thyroid mass (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 21 | 15
Cataract nuclear (Eye disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Ectropion (Eye disorders) | 0 | 1
Entropion (Eye disorders) | 1 | 0
Exfoliation syndrome (Eye disorders) | 1 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal oedema (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 1 | 1
Abdominal compartment syndrome (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 3 | 2
Abdominal incarcerated hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 9
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 2 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 3
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 4 | 6
Colitis ischaemic (Gastrointestinal disorders) | 4 | 2
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 2
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 0
Diverticulum oesophageal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 8
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gallstone ileus (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric hypomotility (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 20 | 33
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 3 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 7 | 19
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 3 | 5
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3
Melaena (Gastrointestinal disorders) | 3 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 4
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Oesophageal motility disorder (Gastrointestinal disorders) | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 3
Pancreatitis acute (Gastrointestinal disorders) | 4 | 3
Pancreatitis relapsing (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal discharge (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 5 | 2
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 12 | 7
Spigelian hernia (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 8
Vomiting (Gastrointestinal disorders) | 3 | 0
Accidental death (General disorders) | 2 | 0
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 8 | 5
Cardiac death (General disorders) | 2 | 1
Catheter site haematoma (General disorders) | 0 | 1
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 23 | 34
Complication associated with device (General disorders) | 0 | 1
Complication of device insertion (General disorders) | 1 | 0
Death (General disorders) | 37 | 32
Device embolisation (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 1
Generalised oedema (General disorders) | 0 | 4
Hernia (General disorders) | 1 | 2
Impaired healing (General disorders) | 1 | 0
Implant site bruising (General disorders) | 1 | 0
Implant site dehiscence (General disorders) | 4 | 1
Implant site dermatitis (General disorders) | 0 | 1
Implant site discharge (General disorders) | 1 | 0
Implant site erosion (General disorders) | 1 | 0
Implant site erythema (General disorders) | 2 | 1
Implant site haematoma (General disorders) | 29 | 25
Implant site haemorrhage (General disorders) | 0 | 3
Implant site irritation (General disorders) | 1 | 0
Implant site pain (General disorders) | 10 | 17
Implant site swelling (General disorders) | 1 | 0
Incarcerated hernia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 1
Mass (General disorders) | 0 | 1
Medical device discomfort (General disorders) | 0 | 1
Medical device site joint pain (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 4 | 5
Non-cardiac chest pain (General disorders) | 13 | 14
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 3 | 0
Pacemaker syndrome (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 1
Phantom shocks (General disorders) | 2 | 4
Polyp (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 5
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 2
Terminal state (General disorders) | 1 | 1
Ulcer (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 0 | 3
Vascular stent thrombosis (General disorders) | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 8 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 9 | 7
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 3
Hepatic congestion (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic lesion (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 2 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 2
Hypersensitivity (Immune system disorders) | 1 | 2
Sarcoidosis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 4 | 2
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 7 | 2
Biliary sepsis (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 11 | 15
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 31 | 41
Chronic sinusitis (Infections and infestations) | 1 | 1
Citrobacter sepsis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 4
Clostridium difficile infection (Infections and infestations) | 3 | 4
Cryptosporidiosis infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 3 | 1
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 6 | 12
Device related sepsis (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 2
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 8 | 11
Emphysematous cholecystitis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 6 | 9
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 1 | 1
Enterococcal infection (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 2 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 3 | 1
Gangrene (Infections and infestations) | 5 | 2
Gastroenteritis (Infections and infestations) | 9 | 5
Gastroenteritis viral (Infections and infestations) | 4 | 3
Gastrointestinal infection (Infections and infestations) | 0 | 1
Graft infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Herpes sepsis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Implant site cellulitis (Infections and infestations) | 2 | 5
Implant site infection (Infections and infestations) | 24 | 44
Incision site cellulitis (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 0 | 3
Infectious colitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 19 | 13
Infusion site infection (Infections and infestations) | 1 | 0
Intestinal sepsis (Infections and infestations) | 2 | 1
Kidney infection (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Labyrinthitis (Infections and infestations) | 1 | 0
Lemierre syndrome (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 2 | 3
Mediastinitis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 3 | 1
Osler's nodes (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 6 | 4
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Parotitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 118 | 112
Pneumonia bacterial (Infections and infestations) | 3 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 2
Pneumonia pseudomonal (Infections and infestations) | 1 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 2
Pneumonia streptococcal (Infections and infestations) | 1 | 1
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 8 | 13
Pyelonephritis (Infections and infestations) | 3 | 2
Pyelonephritis acute (Infections and infestations) | 0 | 3
Pyuria (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 23 | 20
Septic shock (Infections and infestations) | 11 | 9
Staphylococcal bacteraemia (Infections and infestations) | 2 | 4
Staphylococcal infection (Infections and infestations) | 2 | 2
Staphylococcal sepsis (Infections and infestations) | 3 | 3
Stitch abscess (Infections and infestations) | 1 | 0
Stoma site cellulitis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 2 | 1
Syphilis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 2 | 0
Tracheostomy infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 52 | 57
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 15 | 17
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 3 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 2
Wound infection bacterial (Infections and infestations) | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 4 | 7
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 11 | 9
Cardiac vein dissection (Injury, poisoning and procedural complications) | 3 | 1
Cardiac vein perforation (Injury, poisoning and procedural complications) | 1 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 3 | 3
Device deployment issue (Injury, poisoning and procedural complications) | 2 | 2
Device difficult to use (Injury, poisoning and procedural complications) | 1 | 1
Device use issue (Injury, poisoning and procedural complications) | 2 | 1
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 12
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 9 | 7
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 2
Heat exhaustion (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 15 | 11
Humerus fracture (Injury, poisoning and procedural complications) | 3 | 4
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 | 4
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 6 | 5
Limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 3 | 4
Meniscus injury (Injury, poisoning and procedural complications) | 3 | 2
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 2 | 3
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 9 | 5
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pocket erosion (Injury, poisoning and procedural complications) | 3 | 4
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 2 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 2 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 0
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0
Rectal laceration postoperative (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Sacroiliac fracture (Injury, poisoning and procedural complications) | 0 | 1
Scar (Injury, poisoning and procedural complications) | 1 | 0
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Sedation complication (Injury, poisoning and procedural complications) | 1 | 0
Skin scar contracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 3
Splenic rupture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 12 | 11
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 3
Twiddler's syndrome (Injury, poisoning and procedural complications) | 3 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site dissection (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Vena cava injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 2 | 1
Anticoagulation drug level below therapeutic (Investigations) | 1 | 1
Blood glucose decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Cardiac output decreased (Investigations) | 1 | 0
Colonoscopy (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1
Femoral bruit (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 3
Heart rate irregular (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0
Influenza A virus test positive (Investigations) | 0 | 2
International normalised ratio fluctuation (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 1
Pulse absent (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 10 | 12
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 3 | 3
Fluid overload (Metabolism and nutrition disorders) | 3 | 3
Gout (Metabolism and nutrition disorders) | 4 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 8
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 2
Obesity (Metabolism and nutrition disorders) | 5 | 3
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 8 | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 4
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Facial asymmetry (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 34 | 46
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 10
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 12
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 4
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 7
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 1
Ataxia (Nervous system disorders) | 1 | 2
Autonomic nervous system imbalance (Nervous system disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 2 | 1
Carotid artery stenosis (Nervous system disorders) | 5 | 4
Carpal tunnel syndrome (Nervous system disorders) | 3 | 3
Cerebral artery occlusion (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 4
Cerebral infarction (Nervous system disorders) | 2 | 3
Cerebrovascular accident (Nervous system disorders) | 34 | 26
Cognitive disorder (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 5 | 2
Dementia Alzheimer's type (Nervous system disorders) | 3 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 6 | 8
Dizziness postural (Nervous system disorders) | 0 | 2
Dysarthria (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 4 | 4
Facial paralysis (Nervous system disorders) | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 5 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 5 | 2
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial mass (Nervous system disorders) | 1 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Intraneural cyst (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 2 | 11
Lacunar infarction (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 3 | 1
Lumbar radiculopathy (Nervous system disorders) | 2 | 0
Metabolic encephalopathy (Nervous system disorders) | 4 | 1
Migraine (Nervous system disorders) | 1 | 0
Myelomalacia (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Neurodegenerative disorder (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 2
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Polyneuropathy alcoholic (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 4
Restless legs syndrome (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 3 | 4
Seizure like phenomena (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 24 | 28
Thalamic infarction (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 26 | 16
Tremor (Nervous system disorders) | 0 | 2
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 1 | 0
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Device battery issue (Product Issues) | 3 | 1
Device breakage (Product Issues) | 0 | 1
Device capturing issue (Product Issues) | 9 | 9
Device connection issue (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 3 | 4
Device electrical impedance issue (Product Issues) | 5 | 6
Device end of service (Product Issues) | 0 | 1
Device extrusion (Product Issues) | 1 | 5
Device failure (Product Issues) | 0 | 2
Device inappropriate shock delivery (Product Issues) | 6 | 11
Device lead damage (Product Issues) | 19 | 24
Device lead issue (Product Issues) | 7 | 11
Device loosening (Product Issues) | 0 | 1
Device malfunction (Product Issues) | 10 | 14
Device pacing issue (Product Issues) | 16 | 6
Device stimulation issue (Product Issues) | 11 | 20
Implant subsidence (Product Issues) | 0 | 1
Lead dislodgement (Product Issues) | 39 | 37
Oversensing (Product Issues) | 1 | 10
Thrombosis in device (Product Issues) | 1 | 0
Undersensing (Product Issues) | 1 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 1
Intentional self-injury (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 9 | 9
Psychotic disorder (Psychiatric disorders) | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 66 | 72
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 1
Calculus bladder (Renal and urinary disorders) | 3 | 0
Calculus urethral (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 3 | 7
End stage renal disease (Renal and urinary disorders) | 3 | 5
Haematuria (Renal and urinary disorders) | 4 | 5
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Myeloma cast nephropathy (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 5 | 5
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Pulmonary renal syndrome (Renal and urinary disorders) | 1 | 0
Renal aneurysm (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal embolism (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 8 | 11
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 2
Renal mass (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 4 | 6
Urethral disorder (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 5 | 7
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 | 7
Breast mass (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Rectoprostatic fistula (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 2 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 22
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 45 | 32
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 18
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 11
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 30 | 32
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Brow ptosis (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 2
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 | 7
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 1
Elderly (Social circumstances) | 1 | 0
Familial risk factor (Social circumstances) | 1 | 0
Argon plasma coagulation (Surgical and medical procedures) | 0 | 1
Arteriovenous fistula operation (Surgical and medical procedures) | 1 | 0
Blepharoplasty (Surgical and medical procedures) | 1 | 0
Cataract operation (Surgical and medical procedures) | 1 | 1
Coronary artery bypass (Surgical and medical procedures) | 1 | 0
Heart transplant (Surgical and medical procedures) | 0 | 1
Hernia repair (Surgical and medical procedures) | 2 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 1
Jejunostomy (Surgical and medical procedures) | 1 | 0
Leg amputation (Surgical and medical procedures) | 1 | 0
Metatarsal excision (Surgical and medical procedures) | 0 | 1
Mitral valve replacement (Surgical and medical procedures) | 1 | 0
Neurectomy (Surgical and medical procedures) | 1 | 0
Prostatectomy (Surgical and medical procedures) | 0 | 1
Wound treatment (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aneurysm ruptured (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 8 | 7
Aortic dissection (Vascular disorders) | 2 | 3
Aortic rupture (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 8 | 16
Arterial disorder (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 5
Bleeding varicose vein (Vascular disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 1
Brachiocephalic artery occlusion (Vascular disorders) | 0 | 1
Brachiocephalic vein occlusion (Vascular disorders) | 0 | 1
Brachiocephalic vein stenosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 13 | 13
Haematoma (Vascular disorders) | 8 | 3
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 2 | 1
Hypertensive emergency (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 15 | 16
Hypovolaemic shock (Vascular disorders) | 1 | 1
Intermittent claudication (Vascular disorders) | 3 | 1
Ischaemia (Vascular disorders) | 1 | 2
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 5 | 5
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 6
Peripheral artery occlusion (Vascular disorders) | 2 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 3
Peripheral artery thrombosis (Vascular disorders) | 1 | 1
Peripheral embolism (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 9 | 9
Peripheral vascular disorder (Vascular disorders) | 5 | 6
Peripheral venous disease (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 3 | 2
Subclavian vein occlusion (Vascular disorders) | 0 | 2
Subclavian vein stenosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 3 | 0
Varicose vein (Vascular disorders) | 1 | 1
Vasculitis (Vascular disorders) | 0 | 1
Vena cava embolism (Vascular disorders) | 0 | 1
Venous occlusion (Vascular disorders) | 8 | 3
Venous stenosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 2 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TYRX Envelope (N=3495) | Control (N=3488)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac discomfort (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 3
Exercise tolerance decreased (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Impaired healing (General disorders) | 3 | 1
Implant site bruising (General disorders) | 7 | 2
Implant site dehiscence (General disorders) | 4 | 3
Implant site discharge (General disorders) | 3 | 0
Implant site erythema (General disorders) | 4 | 4
Implant site extravasation (General disorders) | 1 | 1
Implant site haematoma (General disorders) | 56 | 43
Implant site haemorrhage (General disorders) | 6 | 5
Implant site inflammation (General disorders) | 1 | 0
Implant site irritation (General disorders) | 4 | 2
Implant site oedema (General disorders) | 1 | 1
Implant site pain (General disorders) | 23 | 20
Implant site pruritus (General disorders) | 3 | 2
Implant site rash (General disorders) | 6 | 0
Implant site scar (General disorders) | 1 | 0
Implant site swelling (General disorders) | 13 | 10
Implant site vesicles (General disorders) | 1 | 1
Medical device site laceration (General disorders) | 0 | 1
Medical device site pain (General disorders) | 1 | 0
Medical device site paraesthesia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pacemaker generated arrhythmia (General disorders) | 1 | 0
Pacemaker syndrome (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 1
Phantom shocks (General disorders) | 4 | 2
Pyrexia (General disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 2
Implant site cellulitis (Infections and infestations) | 2 | 2
Implant site infection (Infections and infestations) | 8 | 14
Infection (Infections and infestations) | 1 | 1
Infusion site cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 5
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Stitch abscess (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Cardiac vein dissection (Injury, poisoning and procedural complications) | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 2 | 5
Incision site haemorrhage (Injury, poisoning and procedural complications) | 3 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Incision site pruritus (Injury, poisoning and procedural complications) | 2 | 0
Incision site vesicles (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 1 | 0
Procedural anxiety (Injury, poisoning and procedural complications) | 0 | 1
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 1
Blood creatinine increased (Investigations) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Device capturing issue (Product Issues) | 4 | 3
Device dislocation (Product Issues) | 2 | 0
Device electrical finding (Product Issues) | 1 | 0
Device electrical impedance issue (Product Issues) | 7 | 4
Device inappropriate shock delivery (Product Issues) | 3 | 3
Device lead damage (Product Issues) | 1 | 1
Device lead issue (Product Issues) | 3 | 3
Device malfunction (Product Issues) | 1 | 0
Device pacing issue (Product Issues) | 7 | 9
Device signal detection issue (Product Issues) | 2 | 0
Device stimulation issue (Product Issues) | 44 | 37
Electromagnetic interference (Product Issues) | 1 | 0
Lead dislodgement (Product Issues) | 2 | 0
Oversensing (Product Issues) | 11 | 10
Undersensing (Product Issues) | 3 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 4
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 2
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 2
Venous occlusion (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after release of a multi-center publication per the publication strategy following Medtronic's review for disclosure of confidential information ("CI"), technical correctness, disclosure of patentable or copyrightable material, and selection and order of publications by the publications committee. Any such CI and/or item identified as not technically correct is deleted prior to publication/presentation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT02277990/Prot_SAP_000.pdf